CLINICAL TRIAL: NCT02248545
Title: Autoimmune Diseases And Serum Anti-Nuclear Antibodies Positivity In Non-Celiac Wheat Sensitivity Patients
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, Principal investigator, University of Palermo
Other Study IDs: ACPM06
Record Dates: First submitted 2014-09-20; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Non-Celiac Wheat Sensitivity
Keywords: Non-Celiac Wheat Sensitivity; Autoimmune diseases; Anti-nuclear antibodies; Celiac disease; Irritable bowel syndrome
MeSH Terms: conditions — Autoimmune Diseases; Celiac Disease; Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Non-celiac Wheat Sensitivity Patients: Consecutive adult patients with irritable bowel syndrome (IBS)-like clinical presentation, according to Rome II criteria, and a definitive diagnosis of NCWS.
- Celiac Disease Patients: Celiac disease adult patients, sex- and age-matched, diagnosed according to standard criteria, during the same study period, chosen at random and enrolled as first control group.
- Irritable Bowel Syndrome Patients: Irritable Bowel Syndrome adult patients, sex- and age-matched, diagnosed according to Rome II criteria, and unrelated to NCWS or other food "intolerance", during the same study period, chosen at random and enrolled as second control group.

SUMMARY:
Celiac disease (CD) is an immune-based reaction to dietary gluten (storage protein for wheat, barley, and rye) that primarily affects the small intestine in genetically predisposed patients and resolves with exclusion of gluten from the diet. Patients with CD show circulating autoantibodies (anti-transglutaminase, anti-tTG) and suffer from the destruction of a specific tissue cell type (the enterocytes) by CD8+ T cells. Furthermore, other autoimmune diseases have been reported in association to CD in 20-30% of the cases. In the last few year, a new clinical entity emerged, which seems include patients who consider themselves to be suffering from problems caused by wheat and/or gluten ingestion, even though they do not have CD or wheat allergy. This clinical condition has been named "Non-Celiac Gluten Sensitivity" (6), but, in a recent paper, the investigators suggested the term "Non-Celiac Wheat Sensitivity" (NCWS), since, to date, it is not known what component of wheat really causes the symptoms. The doubt areas about the NCWS regard also its pathogenesis as, despite some papers evidenced an intestinal immunologic activation, others excluded it. To explore the presence of autoimmunity in NCWS, the investigators evaluated: a) the frequency of autoimmune diseases and b) the frequency of serum anti-nuclear antibodies (ANA) positivity in newly diagnosed NCWS, compared to CD patients.

DETAILED DESCRIPTION:
Celiac disease (CD) is an immune-based reaction to dietary gluten (storage protein for wheat, barley, and rye) that primarily affects the small intestine in genetically predisposed patients and resolves with exclusion of gluten from the diet. Although CD is not surely placed among the autoimmune diseases, patients with CD show circulating autoantibodies (anti-transglutaminase, anti-tTG) and suffer from the destruction of a specific tissue cell type (the enterocytes) by CD8+ T cells. Furthermore, other autoimmune diseases have been reported in association to CD in 20-30% of the cases. In the last few year, a new clinical entity emerged, which seems include patients who consider themselves to be suffering from problems caused by wheat and/or gluten ingestion, even though they do not have CD or wheat allergy. This clinical condition has been named "Non-Celiac Gluten Sensitivity" (6), but, in a recent paper, the investigators suggested the term "Non-Celiac Wheat Sensitivity" (NCWS), since, to date, it is not known what component of wheat really causes the symptoms. The doubt areas about the NCWS regard also its pathogenesis as, despite some papers evidenced an intestinal immunologic activation, others linked NCWS to the dietary FODMAPs (Fermentable Oligo-di and Mono-saccharides, And Polyols) load, thus excluding an immunologic involvement in the NCWS. To explore the presence of autoimmunity in NCWS, in the present study the investigators evaluated: a) the frequency of autoimmune diseases and b) the frequency of serum anti-nuclear antibodies (ANA) positivity in newly diagnosed NCWS and CD patients.

ELIGIBILITY:
Inclusion Criteria:

* To diagnose NCWS the recently proposed criteria were adopted. All the patients met the following criteria
* negative serum anti-transglutaminase (anti-tTG) and anti-endomysium (EmA) IgA and IgG antibodies
* absence of intestinal villous atrophy
* negative IgE-mediated immune-allergy tests to wheat (skin prick tests and/or serum specific IgE detection)
* resolution of the IBS symptoms on standard elimination diet, excluding wheat, cow's milk, egg, tomato, chocolate, and other self-reported food(s) causing symptoms
* symptom reappearance on double-blind placebo-controlled (DBPC) wheat challenge. As we previously described in other studies, DBPC cow's milk protein challenge and other "open" food challenges were performed too.
* Additional inclusion criteria were:
* age >18 years
* follow-up duration longer than six months after the initial diagnosis
* at least two outpatient visits during the follow-up period.

Exclusion Criteria:

* positive EmA in the culture medium of the duodenal biopsies, also in the case of normal villi/crypts ratio in the duodenal mucosa
* self-exclusion of wheat from the diet and refusal to reintroduce it, before entering the study
* other "organic" gastrointestinal disorders
* nervous system disease and/or major psychiatric disorder
* physical impairment limiting physical activity
* menopause
* steroid and sex steroid therapy, hormone replacement therapy or ovariectomy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included consecutive adult patients with irritable bowel syndrome (IBS)-like clinical presentation, according to Rome II criteria, and a definitive diagnosis of NCWS, referred at the Internal Medicine Department of the University Hospital of Palermo, Italy, and at the Internal Medicine Department of the Hospital of Sciacca, Agrigento, Italy, between July 2011 and July 2013.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2011-07; Primary Completion 2013-07 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Organ- and non-organ specific autoantibodies | At first visit
  We evaluated, by ELISA and Immunofluorescence, organ- and non-organ specific autoantibodies, i.e. Anti-Nuclear Antibodies (ANA) IgG, anti double-strand (anti-ds) DNA IgG Antibodies, Anti-Mitochondrial Antibodies (AMA), Liver Kidney Microsome (LKM) IgG Antibodies, Anti-Smooth Muscle Antibodies (ASMA) IgG, anti-Sjogren's Syndrome antigen A (anti-SSA) IgG Antibodies, anti-Sjogren's Syndrome antigen B (anti-SSB) IgG Antibodies, anti-Smith (anti-Sm) IgG Antibodies, anti-ThyroPerOxidase (anti-TPO) IgG Antibodies, anti-ThyroGlobulin (anti-TG) IgG Antibodies, anti-Glutamic Acid Decarboxylase (anti-GAD) IgG Antobodies, and Islet Cell Antibodies (ICA) IgG.

SECONDARY OUTCOMES:
Questionnaire for autoimmunity. | At first visit
  The presence of autoimmune disorders was evaluated by a structured questionnaire, with the assistance of ad hoc-trained personnel, and review of patient' clinical records. The presence of one of the following diseases was looked for in all subjects: connective tissue diseases, autoimmune endocrinological diseases, autoimmune hepatitis, primary biliary cirrhosis, epilepsy with cerebral calcification, unexplained cerebellar ataxia, alopecia, psoriasis, dermatitis herpetiform, atrophic autoimmune gastritis, and immune anemia, neutropenia, or thrombocytopenia. The hospital records of all patients diagnosed for an autoimmune disorder were thoroughly examined to verify whether the recognized diagnostic criteria for each disorder had been fulfilled, together with age at diagnosis of the diseases and treatment received.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, MD, PhD, Principal Investigator — Internal Medicine Department of the Hospital of Sciacca (Agrigento)
Locations (3):
- Italy (3):
  - Internal Medicine Department of the Hospital of Sciacca (Agrigento), Sciacca, Agrigento
  - Gastroenterology Unit of the "Civico" Hospital of Palermo, Palermo, Palermo
  - Internal Medicine Department of the University Hospital of Palermo, Palermo, Palermo

REFERENCES:
- [Result] Rubio-Tapia A, Hill ID, Kelly CP, Calderwood AH, Murray JA; American College of Gastroenterology. ACG clinical guidelines: diagnosis and management of celiac disease. Am J Gastroenterol. 2013 May;108(5):656-76; quiz 677. doi: 10.1038/ajg.2013.79. Epub 2013 Apr 23. PMID 23609613
- [Result] Sollid LM, Jabri B. Triggers and drivers of autoimmunity: lessons from coeliac disease. Nat Rev Immunol. 2013 Apr;13(4):294-302. doi: 10.1038/nri3407. Epub 2013 Mar 15. PMID 23493116
- [Result] Sategna Guidetti C, Solerio E, Scaglione N, Aimo G, Mengozzi G. Duration of gluten exposure in adult coeliac disease does not correlate with the risk for autoimmune disorders. Gut. 2001 Oct;49(4):502-5. doi: 10.1136/gut.49.4.502. PMID 11559646
- [Result] Biagi F, Pezzimenti D, Campanella J, Corazza GR. Gluten exposure and risk of autoimmune disorders. Gut. 2002 Jul;51(1):140-1. doi: 10.1136/gut.51.1.140-a. No abstract available. PMID 12077109
- [Result] Verdu EF, Armstrong D, Murray JA. Between celiac disease and irritable bowel syndrome: the "no man's land" of gluten sensitivity. Am J Gastroenterol. 2009 Jun;104(6):1587-94. doi: 10.1038/ajg.2009.188. PMID 19455131
- [Result] Catassi C, Bai JC, Bonaz B, Bouma G, Calabro A, Carroccio A, Castillejo G, Ciacci C, Cristofori F, Dolinsek J, Francavilla R, Elli L, Green P, Holtmeier W, Koehler P, Koletzko S, Meinhold C, Sanders D, Schumann M, Schuppan D, Ullrich R, Vecsei A, Volta U, Zevallos V, Sapone A, Fasano A. Non-Celiac Gluten sensitivity: the new frontier of gluten related disorders. Nutrients. 2013 Sep 26;5(10):3839-53. doi: 10.3390/nu5103839. PMID 24077239
- [Result] Carroccio A, Rini G, Mansueto P. Non-celiac wheat sensitivity is a more appropriate label than non-celiac gluten sensitivity. Gastroenterology. 2014 Jan;146(1):320-1. doi: 10.1053/j.gastro.2013.08.061. Epub 2013 Nov 22. No abstract available. PMID 24275240
- [Derived] Mansueto P, Soresi M, Candore G, Garlisi C, Fayer F, Gambino CM, La Blasca F, Seidita A, D'Alcamo A, Lo Sasso B, Florena AM, Geraci G, Caio G, Volta U, De Giorgio R, Ciaccio M, Carroccio A. Autoimmunity Features in Patients With Non-Celiac Wheat Sensitivity. Am J Gastroenterol. 2021 May 1;116(5):1015-1023. doi: 10.14309/ajg.0000000000000919. PMID 33009065